CLINICAL TRIAL: NCT04768842
Title: Comparative Pharmacokinetics of LY3209590 After Administration of a Lyophilized Formulation and a Solution Formulation in Healthy Participants
Brief Title: A Study of Two Different Formulations of LY3209590 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16494; I8H-MC-BDCJ (Other: Eli Lilly and Company); 2020-003738-19 (EudraCT Number)
Record Dates: First submitted 2021-02-23; First posted 2021-02-24 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09-15

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3209590 Lyophilized Formulation (Experimental): LY3209590 as lyophilized formulation administered subcutaneously (SC) in one of the two study periods.
  Interventions: Drug: LY3209590
- LY3209590 Solution Formulation (Experimental): LY3209590 as solution formulation administered SC in one of the two study periods.
  Interventions: Drug: LY3209590

INTERVENTIONS:
Drug: LY3209590 — Administered SC.

SUMMARY:
The main purpose of this study is to look at the amount of the study drug, LY3209590, that gets into the blood stream and how long it takes the body to get rid of LY3209590 when given as different formulations. The tolerability of LY3209590 will also be evaluated and information about any side effects experienced will be collected. The study will last up to 142 days.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or non-pregnant females. Additionally, women of childbearing potential must test negative for pregnancy
* Have a body mass index (BMI) of 18 to 35 kilograms per square meter (kg/m²), inclusive at screening
* Have blood pressure, pulse rate, blood and urine laboratory test results that are acceptable for the study
* Have veins suitable for blood sampling
* Have given written informed consent approved by Lilly and the ethical review board governing the site

Exclusion Criteria:

* Have or used to have health problems that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Are women who are pregnant or lactating
* Have a history of multiple and/or severe allergic reactions
* Show clinical evidence of HIV, hepatitis C, or hepatitis B, and/or test positive
* Regularly use known drugs of abuse or with positive drug results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3209590 | Predose on Day 1 through Day 65
  PK: Cmax of LY3209590
PK: Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC[0-inf]) of LY3209590 | Predose on Day 1 through Day 65
  PK: AUC(0-inf) of LY3209590

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No